CLINICAL TRIAL: NCT00351663
Title: Prospective Randomised Study of the Effect of Vasopressors on the Anti Xa Response to Enoxaparin in Critically Ill Patients
Brief Title: The Effect of Vasopressors on the Anti Xa Response to Enoxaparin in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr Sharon Einav, Dr., Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: einav-1-ctil
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Venous Thrombosis; Critical Illness
Keywords: Venous Thrombosis; Critical Illness; Blood Coagulation; Factor Xa
MeSH Terms: conditions — Venous Thrombosis; Critical Illness; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV by weight (Active Comparator): intravenous dose of 0.5 mg/kg enoxaparin once daily
  Interventions: Drug: Enoxaparine
- SC fixed dose (Active Comparator): subcutaneous fixed dose of 40 mg enoxaparin once daily
  Interventions: Drug: Enoxaparine
- SC by weight (Active Comparator): subcutaneous dose of 0.5 mg/kg enoxaparin once daily
  Interventions: Drug: Enoxaparine

INTERVENTIONS:
Drug: Enoxaparine — Patients considered eligible will be divided into 2 groups- those receiving vasopressor support and those not receiving vasopressor support at the time of inclusion. The patients in each group will be randomized to receive enoxaparin in accordance with one of the following DVT prophylaxis protocols:
  1. Intravenous Enoxaparine according to their weight (0.5mg/kg x 1/day)
  2. Subcutaneous Enoxaparine according to their weight (0.5mg/kg x 1/day)
  3. Subcutaneous Enoxaparine 40mg x1/day

SUMMARY:
The purpose of this study is to evaluate the efficacy of 3 different dosing regimens of enoxaparin in achieving adequate antithrombotic aFXa levels in critically ill patients.

The relationship between appearance of DVT and antithrombotic aFXa levels will also be assessed and risk factors associated with inadequate aFXa levels under standard enoxaparin dosages will be searched for.

DETAILED DESCRIPTION:
Critically ill patients are at increased risk of venous thrombosis and embolism from DVT. Low molecular weigh heparins such as enoxaparin (clexane) have more favorable pharmacokinetic/ pharmacodynamic profiles, equivalent or improved efficacy (e.g. in post trauma and orthopedic surgery patients) and fewer bleeding complications than low-dose unfractionated heparin. These medications are currently recommended for DVT prophylaxis in critically ill patients and are usually administered subcutaneously (SQ). The antithrombotic activity of LMWHs correlates with peak aFXa levels. However, the the appropriate dose and dosing interval of enoxaparin for DVT prophylaxis in critically ill surgical patients has not been established and in particular remains unknown for those patients with severe peripheral edema ans/or decreased peripheral circulation due to therapy with vasopressors. Several studies have recently demonstrated questionable efficacy of standard daily enoxaparin dosing for critically ill patients as DVT prophylaxis.

The current study will be a prospective, randomized, cohort study, conducted at the Shaare Zedek Medical Center over a period of 1 year (100 patients). All critically ill patients aged ≥18 years with a predicted requirement of mechanical ventilation for >3 days will be included. Data collection will be performed anonymously and will include patient demographics and admission details, duplex monitoring for DVT and daily recording of APACHE II scores, renal function, coagulation profile and overall dose of vasopressors.

Patients will be randomized to receive enoxaparin in accordance three DVT prophylaxis protocols- IV by weight, SQ by weight or SQ 40mg x1/day (standard). Blood samples for the evaluation of aFXa will be drawn twice daily for peak and trough activity over a period of 5 days. No further changes will be made in the standard therapy. Patient outcomes and occurrence of adverse events will be recorded. The principle outcome variable will be achievement of target peak and trough levels of aFXa during the 5 day study period.

ELIGIBILITY:
Inclusion Criteria:

All critically ill patients, aged ≥18 years, with a predicted requirement for mechanical ventilation of more than 3 days and for whom venous thromboembolic prophylaxis is indicated.

-

Exclusion Criteria:

1. Patients requiring full anticoagulation
2. Administration of unfractionated heparin in the 8hrs preceding study entry
3. Existing contraindication to prophylactic dose of enoxaparin.
4. Platelets < 75,000
5. Significant renal failure (creatinine clearance <30 ml/min/m2) [39]
6. BMI > 30
7. INR > 1.7
8. Any conditions precluding treatment in the opinion of the primary physician
9. Patient /surrogate refusal

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-02; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of the dosing protocols of enoxaparin for critically ill patients on aFXa activity | 5 days

SECONDARY OUTCOMES:
bleeding/thrombotic complications | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Einav-Bromiker, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Result] Helviz Y, Dzigivker I, Raveh-Brawer D, Hersch M, Zevin S, Einav S. Anti-Factor Xa Activity of Prophylactic Enoxaparin Regimens in Critically Ill Patients. Isr Med Assoc J. 2016 Feb;18(2):108-13. PMID 26979004